CLINICAL TRIAL: NCT02265172
Title: Does Orthopaedic Manual Therapy Assessment of Patients Referred to Orthopaedic Surgeon Bring Any Changes to Referral Routines, Patient Satisfaction and Health-related Variables?
Brief Title: Physiotherapy Assessment of Patients Referred to Orthopaedic Surgeon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EPN GBG 328-09
Record Dates: First submitted 2014-10-06; First posted 2014-10-15 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-09

CONDITIONS: Musculoskeletal Pain
Keywords: Physiotherapy; Orthopaedic; Primary care
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy screening (Experimental): Screening consisted of a 60-min appointment including assessment, diagnosis and management. The patients received advice regarding ergonomics, exercises and/or treatment when needed. Management options were;
  * Referral for orthopaedic surgeon consultation.
  * Referral back to the patient's General Practitioner.
  * Referral for further investigation.
  * Referral to the physiotherapy or the occupational therapy clinic.
  Interventions: Procedure: Physiotherapy screening
- Standard practice (orthopaedic surgeon) (Active Comparator): Appointment was 15 min, including assessment, diagnosis and management. The patients received advice, prescriptions or injections when needed. Management options were;
  * Referral for orthopaedic intervention.
  * Referral back to the patient's General Practitioner.
  * Referral for further investigation.
  * Referral to the physiotherapy or the occupational therapy clinic.
  Interventions: Procedure: Standard practice

INTERVENTIONS:
Procedure: Physiotherapy screening — Physiotherapy screening.
  Arms: Physiotherapy screening
Procedure: Standard practice — Orthopaedic surgeon assessment
  Arms: Standard practice (orthopaedic surgeon)

SUMMARY:
Many patients with musculoskeletal pain in primary healthcare are referred to orthopaedic surgeon, however, a relatively low percentage of these patients are considered suitable for orthopaedic intervention.

Physiotherapists are suitable for musculoskeletal assessments and are used as such in many countries i.e. Advanced Practice Physiotherapists or Extended Scope Physiotherapists, however, this is not an existing model of care in Sweden. To be able to consider this model for implementation in Sweden it is necessary to evaluate it from a healthcare as well as from a patient perspective.

The study is a randomised controlled trial. Overall aim is to evaluate if a orthopaedic manual therapy assessment (physiotherapy) assessment of patients referred to orthopaedic surgeon bring any changes to referral routines, patient satisfaction and health-related variables when compared to standard practice.

DETAILED DESCRIPTION:
The study is a randomised controlled trial. Overall aim is to evaluate if a orthopaedic manual therapy assessment (physiotherapy) assessment of patients referred to orthopaedic surgeon bring any changes to referral routines, patient satisfaction and health-related variables when compared to standard practice. Patients were randomised to either physiotherapy assessment or standard practice (orthopaedic surgeon assessment).

ELIGIBILITY:
Inclusion Criteria:

* patients referred for orthopaedic surgeon with sub acute (four weeks to three months) or chronic (>three months) musculoskeletal pain who had the ability to understand written and spoken Swedish.

Exclusion Criteria:

* diagnosed hallux valgus, ganglion or trigger finger.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of referrals after consultation as a measure of Management outcome | 12 months

SECONDARY OUTCOMES:
Scores on the questionnaire Quality from the Patient Perspective as a measure of Patient satisfaction | 30 days
Scores on the EuroQol-5D as a measure of Health-related quality of life | 12 months
Scores on the Pain Disability Index as a measure of Pain-related disability | 12 months
Number of sick-leave days | 12 months
Cost per quality adjusted life year (QUALY) gained as a measure of cost-utitily | 12 months
  QUALYs are calculated from the EuroQol-5D
Scores on the Pain Belief Screening Instrument as a measure of risk for long-term disability | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Larsson, PhD, Study Director — Närhalsan Research and development, Region of Västra Götaland

REFERENCES:
- [Result] Samsson K, Larsson ME. Physiotherapy screening of patients referred for orthopaedic consultation in primary healthcare - a randomised controlled trial. Man Ther. 2014 Oct;19(5):386-91. doi: 10.1016/j.math.2013.10.004. Epub 2013 Oct 29. PMID 24246908
- [Result] Samsson KS, Larsson ME. Physiotherapy triage assessment of patients referred for orthopaedic consultation - Long-term follow-up of health-related quality of life, pain-related disability and sick leave. Man Ther. 2015 Feb;20(1):38-45. doi: 10.1016/j.math.2014.06.009. Epub 2014 Jul 15. PMID 25088308
- [Derived] Samsson KS, Bernhardsson S, Sandborgh M, Larsson MEH. The association between screened psychological risk for disability and appropriateness of orthopedic surgery in patients with musculoskeletal disorders - data from a Swedish RCT in primary care 2009-2011. Physiother Theory Pract. 2025 Aug;41(8):1579-1586. doi: 10.1080/09593985.2024.2448709. Epub 2025 Jan 5. PMID 39757368
- [Derived] Samsson KS, Bernhardsson S, Larsson ME. Perceived quality of physiotherapist-led orthopaedic triage compared with standard practice in primary care: a randomised controlled trial. BMC Musculoskelet Disord. 2016 Jun 10;17:257. doi: 10.1186/s12891-016-1112-x. PMID 27286829